CLINICAL TRIAL: NCT07331155
Title: An Open-label, Multicenter, Phase II Clinical Study to Evaluate the Efficacy and Safety of LBL-024 in Combination With Other Drugs for the Treatment of Patients With Advanced Solid Tumour[Substudy Number 03(ESCC)]
Brief Title: A Phase II Clinical Study of LBL-024 Combination Therapy in Patients With Advanced Solid Tumour[Substudy 03(ESCC)]
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanjing Leads Biolabs Co.,Ltd (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBL-024-CN004_03(ESCC)
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumour
MeSH Terms: interventions — Injections; Cisplatin; Paclitaxel; tislelizumab; Fluorouracil; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBL-024+Paclitaxel+Cisplatin/LBL-024+5-Fluorouracil/capecitabine + cisplatin (Experimental): LBL-024+Paclitaxel+Cisplatin/LBL-024+5-Fluorouracil/capecitabine + cisplatin.
  Capecitabine is orally administered and other drugs are Intravenous infusion.
  Interventions: Drug: LBL-024 for Injection; Drug: Cisplatin Injection; Drug: Paclitaxel Injection; Drug: 5-Fluorouracil injection; Drug: Capecitabine tablets
- Tislelizumab+Paclitaxel+Cisplatin/Tislelizumab+5-Fluorouracil/capecitabine + cisplatin (Active Comparator): Tislelizumab+Paclitaxel+Cisplatin/Tislelizumab+5-Fluorouracil/capecitabine + cisplatin.
  Capecitabine is orally administered and other drugs are Intravenous infusion.
  Interventions: Drug: Cisplatin Injection; Drug: Paclitaxel Injection; Drug: Tislelizumab Injection; Drug: 5-Fluorouracil injection; Drug: Capecitabine tablets

INTERVENTIONS:
Drug: LBL-024 for Injection — Intravenous infusion
  Other Names: LBL-024
  Arms: LBL-024+Paclitaxel+Cisplatin/LBL-024+5-Fluorouracil/capecitabine + cisplatin
Drug: Cisplatin Injection — Intravenous infusion
  Other Names: Cisplatin
Drug: Paclitaxel Injection — Intravenous infusion
  Other Names: Paclitaxel
Drug: Tislelizumab Injection — Intravenous infusion
  Other Names: Tislelizumab
  Arms: Tislelizumab+Paclitaxel+Cisplatin/Tislelizumab+5-Fluorouracil/capecitabine + cisplatin
Drug: 5-Fluorouracil injection — Intravenous infusion
  Other Names: 5-Fluorouracil
Drug: Capecitabine tablets — Oral administration
  Other Names: Capecitabine

SUMMARY:
An Open-label, Multicenter, Phase II Clinical Study to Evaluate the Efficacy and Safety of LBL-024 in Combination With Other Drugs for the Treatment of Patients With Advanced Solid Tumour.

DETAILED DESCRIPTION:
This trial is an open-label, multicenter, phase II clinical study of LBL-024 in combination with other drugs for the treatment of patients with advanced oesophageal squamous cell carcinoma (ESCC),to evaluate the efficacy and safety of LBL-024 combination therapy.

This study will have a safety run-in period in which a small number of subjects will be enrolled to receive LBL-024 combination therapy.After the subjects completed the 21-day safety observation, the sponsor and investigator jointly assessed the safety and tolerability of the combination drugs. If safety and tolerability are good, the extension study of combination administration will be continued, the subjects will be continued to be enrolled, and the randomized, open, positive control trial design will be adopted.Subjects who meet the criteria will be randomly assigned to the experimental group and the control group in a ratio of 2: 1.

This trial will enroll up to 110 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the trial treatment regimen, visit schedule, laboratory test, and other requirements of the protocol, and voluntarily enroll in the study and sign the written informed consent.
2. Age ≥ 18 years at the time of signing the informed consent.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
4. The expected survival time is at least 12 weeks.
5. According to the evaluation of RECIST 1.1 standard, the subjects enrolled have at least one measurable lesion.
6. There is adequate organ and bone marrow function,Conforms to laboratory test results.
7. Males with fertility and females of childbearing age are willing to take effective contraceptive measures From the signing of the informed consent form to within 6 months after the last administration of the trial drug (including abstinence, intrauterine device, various hormonal contraception, correct use of contraception Sets，etc）; Women of childbearing age include pre-menopausal women and women within 2 years after menopause. Women of childbearing age must have a negative pregnancy test within 7 days before the first trial drug is administered.

Exclusion Criteria:

1. Participation in clinical studies of antineoplastic agents within 4 weeks before the first use of study drug,or is expected to receive any other form of systemic or local anti-tumor therapy outside the protocol during the study.
2. Use of immunomodulatory drugs within 2 weeks before the first use of study drug,Including but not limited to thymopeptide, interleukins, interferon, etc.
3. Patients with active, or who have had and have the possibility of recurrence of autoimmune diseases.
4. Patients with clinically uncontrollable pleural effusion, pericardial effusion, ascites, and those requiring repeated drainage or medical intervention.
5. The patient has a Medical history of immunodeficiency, including HIV antibody positive.
6. Active hepatitis B or active hepatitis C.
7. Women during pregnancy or lactation.
8. The investigator believes that the subject has other conditions that may affect compliance or are not suitable for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-12-26 (Estimated); Study Completion 2028-12-26 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  Objective Response Rate (complete response (CR) + partial response (PR)), as assessed by Response Evaluation Criteria in Solid Tumors (RECIST 1.1), refers to the percentage of study subjects who achieve a complete response or partial response.

SECONDARY OUTCOMES:
Disease Control Rate(DCR） | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  Percentage of participants achieving CR and PR and stable disease (SD).
Duration of Response(DOR） | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  The period from the participants first achieving CR or PR to disease progression.
Cmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  Maximum serum concentration
Tmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  After taking a single dose, Time to reach maximum plasma concentration
immunogenicity | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  The immunogenicity is evaluated by the incidence of anti-drug antibodies (ADA) and neutralizing antibodies (if applicable) in subjects

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (7):
- China (7):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - AnYang Tumor Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Shandong Cancer Hospital, Jinan, Shandong
  - Suining Central Hospital, Suining, Sichuan

IPD SHARING:
Plan to Share IPD: No